CLINICAL TRIAL: NCT03356119
Title: A Prospective, Single-centre, Non-comparative Feasibility Investigation to Evaluate Performance and Safety of RemovAid ™ Retrieval Device When Used for Removal of Palpable Subdermal Contraceptive Rod Implants.
Brief Title: Pilot Removal of Palpable Subdermal Contraceptive Rod Implants
Acronym: REVALID02
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Inufficient IMD supply due to manufacturing issue
Sponsor: RemovAid AS (Industry)
Collaborators: Karolinska University Hospital (Other); Bill and Melinda Gates Foundation (Other); The Research Council of Norway (Other); Amano Clinical Consulting AB (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: REVALID02
Record Dates: First submitted 2017-11-20; First posted 2017-11-29 (Actual); Last update posted 2018-10-18 (Actual); Status verified 2018-10

CONDITIONS: Removal of Contraceptive Implant
Keywords: Contraceptive Implant

STUDY DESIGN:
Intervention Model Description: All recruited subjects will be assigned to implant removal using the RemovAid IMD. There is no formal comparator in this study. The investigators are investigating design functionality and safety.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- RemovAid arm (Experimental): New IMD Subjects with contraceptive implants to be removed, are subjected to the novel device by personnel skilled in traditional removal.
  Interventions: Device: RemovAid device

INTERVENTIONS:
Device: RemovAid device — The contraceptive implants of the subjects in this arm are removed by the new IMD.

SUMMARY:
There are no implant removal devices on the market by any manufacturer. Overall, the RemovAid™ combines the features of fixation, incision and extraction. This combination of functions has not previously been combined in a single device.

The investigators wish to perform this pilot clinical investigation with the aim to demonstrate that the Investigational Medical Device (IMD), RemovAid ™, may safely and effectively facilitate implant removal. Other aims are to show that the IMD have the potential to reduce procedure length variability, reduce procedural complexity and reduce the need for additional procedural equipment related to CI removal procedures, without causing any harm to the subject.

DETAILED DESCRIPTION:
Detailed Description:

Contraceptive Implants (CIs) were introduced to the commercial market in the early 1980s. They are advocated as a safe and effective method of contraception, and are included on the WHO's Essential Medicines list.

CI manufacturers have focused intense efforts on making insertion of CIs easier, but have largely left CI removals untouched and at the mercy of the various service providers. Different introducers and trocars are available for use with the different CI systems available internationally, and a second generation, single-use trocar is supplied with the Nexplanon® implant system available in Sweden. This second generation trocar has reduced the number of misplaced or deeply inserted CIs, and underlines the benefits of standardizing minor surgical procedures through the use of dedicated medical devices.

The CI removal procedure recommendations have remained essentially unchanged for 40 years, relying on scalpels, forceps and general surgical skills from the service provider. Currently, no standardized technique for removal of CIs exists, and no dedicated CI removal device is found on the commercial market.

Removal of palpable subdermal implants is generally a simple, minor surgical office procedure. However, the procedure for implant removal requires more training and skill than the procedure for insertion. There is a risk of slippage of the scalpel blade or a sudden movement by the client causing inadvertent deeper penetration, in which case any underlying structure could be affected.

Mean removal times, from time of incision until removal of the rod, are consistently reported as less than four minutes, however with ranges from 0.2 - 60 minutes.

Available research shows that the procedure length of the current CI removal procedure is highly variable and reliant on individual operator skills.

ELIGIBILITY:
Inclusion Criteria:

* Female age 18 or older
* Willing to remove a palpable subdermal Implanon/ Nexplanon CI
* Willing and able to give written informed consent for participation in the investigation
* Willing to provide follow-up information according to the Clinical Investigators brochure

Exclusion Criteria:

* Known allergy to local anaesthetic (lidocaine/lignocaine) or disinfectant (chlorhexidine).
* Active skin lesion over the CI.
* The Investigator considers the subject unlikely to comply with investigational procedures, restrictions and requirements.
* Any contraindication for removal of the PI, as judged by the Investigator.
* Any disorders or medications that might affect coagulation, as judged by the Investigator.
* Any conditions suspected to affect healing or increase risk of infection (e.g. keloid tendency, diabetes or any upper arm dermatological condition that may affect upper arm healing)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Only females use contraceptive implants.
Enrollment: 19 (Actual)
Dates: Start 2017-12-12 (Actual); Primary Completion 2018-05-01 (Actual); Study Completion 2018-09-04 (Actual)

PRIMARY OUTCOMES:
Successful removal of implant . | 15 minutes
  Percentage of fixated implants that were successfully removed without the use of additional tools

SECONDARY OUTCOMES:
Frequency, severity, causality and outcome of adverse events (AEs) | 1 week
  Both Anticipated and unanticipated AEs will be recorded, both immediately following the intervention and at follow-up.
Pain during procedure | 5 minutes
  Mean pain score (maximum pain intensity during the procedure) indicated by the subject on a Visual Analogue Scale (VAS) 0-100 mm ruler, assuming that anaesthesia has been properly administered.
Success of fixation of implant | 5 minutes
  Percentage of palpable implants where the implant could be seen and/or felt on both sides of the clamp after maximum three attempts of fixation
Duration of procedure | 25 minutes
  Mean time from making incision until implant is removed. first handling the device until closing the wound.
Technical functionality of device determined by an operators questionnaire | 5 minutes
  Fulfilment of pre-defined technical requirements, as documented on an operator functionality questionnaire. The questionnaire consists of a range of yes/no questions to device functionality
Operators impression of the device | 5 minutes
  The operator's global impression of the IMD will be assessed using a 5-point scale, where 5 is excellent
Subject satisfaction | Time Frame: 5 minutes
  The subject's global assessment of satisfaction with the procedure will be assessed using a 5- point scale, where 5 is excellent

CONTACTS AND LOCATIONS:
Locations (1):
- Karolinska University Hospital, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Committee on Adolescent Health Care Long-Acting Reversible Contraception Working Group, The American College of Obstetricians and Gynecologists. Committee opinion no. 539: adolescents and long-acting reversible contraception: implants and intrauterine devices. Obstet Gynecol. 2012 Oct;120(4):983-8. doi: 10.1097/AOG.0b013e3182723b7d. PMID 22996129
- [Background] Mansour D, Mommers E, Teede H, Sollie-Eriksen B, Graesslin O, Ahrendt HJ, Gemzell-Danielsson K. Clinician satisfaction and insertion characteristics of a new applicator to insert radiopaque Implanon: an open-label, noncontrolled, multicenter trial. Contraception. 2010 Sep;82(3):243-9. doi: 10.1016/j.contraception.2010.04.007. Epub 2010 May 18. PMID 20705152
- [Background] Mommers E, Blum GF, Gent TG, Peters KP, Sordal TS, Marintcheva-Petrova M. Nexplanon, a radiopaque etonogestrel implant in combination with a next-generation applicator: 3-year results of a noncomparative multicenter trial. Am J Obstet Gynecol. 2012 Nov;207(5):388.e1-6. doi: 10.1016/j.ajog.2012.08.002. Epub 2012 Aug 10. PMID 22939402
- [Background] Webb AM. Why go to Tiger Country? A report of two cases of Implanon removal. J Fam Plann Reprod Health Care. 2006 Jul;32(3):193-4. doi: 10.1783/147118906777888233. No abstract available. PMID 16857083
- [Background] Levine JP, Sinofsky FE, Christ MF; Implanon US Study Group. Assessment of Implanon insertion and removal. Contraception. 2008 Nov;78(5):409-17. doi: 10.1016/j.contraception.2008.06.016. Epub 2008 Sep 18. PMID 18929739
- [Background] Funk S, Miller MM, Mishell DR Jr, Archer DF, Poindexter A, Schmidt J, Zampaglione E; Implanon US Study Group. Safety and efficacy of Implanon, a single-rod implantable contraceptive containing etonogestrel. Contraception. 2005 May;71(5):319-26. doi: 10.1016/j.contraception.2004.11.007. PMID 15854630
- See also: World Health Organization. 2014 — http://www.who.int/medicines/publications/essentialmedicines/en/